CLINICAL TRIAL: NCT06021158
Title: A Randomized, Crossover, Pilot Trial to Compare Automated Lyumjev Delivery With Carbohydrate Counting, Qualitative Meal-size Estimation, and Meal Detection in Type 1 Diabetes
Brief Title: A Trial to Compare Automated Lyumjev Delivery With Carbohydrate Counting, Qualitative Meal-size Estimation, and Meal Detection in Type 1 Diabetes
Acronym: Lilly-MEALS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Michael Tsoukas, Associate Professor, Endocrinology & Metabolism, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2024-9583
Record Dates: First submitted 2023-08-24; First posted 2023-09-01 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 1; Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- AID-count (Active Comparator)
  Interventions: Combination Product: Hybrid automated Lyumjev delivery system with carbohydrate counting
- AID-estimate (Experimental)
  Interventions: Combination Product: Hybrid automated Lyumjev delivery system with meal size estimation
- AID-detect (Experimental)
  Interventions: Combination Product: Fully automated Lyumjev delivery system with meal detection

INTERVENTIONS:
Combination Product: Hybrid automated Lyumjev delivery system with carbohydrate counting — In this system, a Lyumjev insulin bolus is initiated at mealtime based on the total grams of carbohydrates counted. This is the same as commercial hybrid closed-loop insulin therapy (standard treatment).
  Arms: AID-count
Combination Product: Hybrid automated Lyumjev delivery system with meal size estimation — In this system, a Lyumjev insulin bolus is initiated at mealtime based on the qualitative amount of carbohydrates estimated (e.g., low-carb meal).
  Arms: AID-estimate
Combination Product: Fully automated Lyumjev delivery system with meal detection — In this system, the patient does not initiate a Lyumjev insulin bolus at mealtime. An algorithm is used to detect a meal and administer a subsequent bolus, rather than requiring a carbohydrate count.
  Arms: AID-detect

SUMMARY:
The goal of this pilot trial is to compare three meal strategies using an ultra-rapid insulin (Lyumjev) and an automated insulin delivery system. The meal strategies to be investigated are carbohydrate counting, qualitative meal announcement (e.g., low-carb meal), and meal detection. The investigators are doing this research to evaluate if carbohydrate counting can be simplified in patients with type 1 diabetes.

Participants will test each meal strategy in random order, and each meal strategy will be 21 days long. For the duration of each meal strategy, participants will use an automated insulin delivery system or "artificial pancreas" with an ultra-rapid insulin called Lyumjev.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes for at least 12 months. The diagnosis of type 1 diabetes is based on the investigator's judgment per local and international guideline criteria.
* Insulin pump use for at least 3 months.
* Individuals of childbearing potential must agree to use a highly effective method of birth control.
* Willing to switch to Lyumjev insulin for the duration of the study.

Exclusion Criteria:

* Use of oral antihyperglycemic agents within 2 weeks of admission (SGLT2i, metformin…); 1 month for GLP1-RA.
* Use of glucocorticoids (except low, stable doses and inhaled steroids).
* Use of hydroxyurea.
* Planned or ongoing pregnancy.
* Breastfeeding.
* Diabetic ketoacidosis and/or severe hypoglycemia episode (defined as requiring the assistance of another person, due to altered consciousness, to administer carbohydrates, glucagon, or other resuscitative actions) within one month of admission.
* Clinically significant retinopathy, nephropathy, or neuropathy as judged by the investigator.
* Recent (<6 months) acute macrovascular event e.g., acute coronary syndrome or cardiac surgery.
* Known hypersensitivity to the study drug or its excipients.
* Other serious medical illness likely to interfere with study participation or with the ability to complete the trial, as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of time of glucose levels spent in the target range (3.9-10.0 mmol/L) | 14 days

SECONDARY OUTCOMES:
Percentage of time of glucose levels spent in the following ranges: - between 3.9 and 7.8 mmol/L - below 3.9 mmol/L - below 3.0 mmol/L - above 10.0 mmol/L - above 13.9 mmol/L | 14 days
Mean glucose levels | 14 days
Standard deviation of glucose levels | 14 days
Standard deviation of insulin delivery | 14 days
Coefficient of variance of glucose levels | 14 days
Coefficient of variance of insulin delivery | 14 days
Total insulin delivery (overall, basal, and bolus) | 14 days
Area under the sensor glucose concentration-time curve (AUC) from 0-1 hours, 0-2 hours, 0-3 hours, 0-4 hours, and 0-5 hours after meal insulin boluses | 14 days
Area under the sensor glucose concentration-time curve (AUC) from 1-2 hours, 2-3 hours, 3-4 hours, and 4-5 hours after meal insulin boluses | 14 days
Decremental sensor glucose concentration for the duration of announced exercise periods | 14 days
Area under the sensor glucose concentration-time curve (AUC) from 0-1 hours, 0-2 hours, 0-3 hours, 0-4 hours, and 0-5 hours after the end of announced exercise periods | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tsoukas, M.D., Principal Investigator — Royal Victoria Hospital, Belfast; Ahmad Haidar, Ph.D., Study Chair — Research Institute of the McGill University University Health Centre; Laurent Legault, M.D., Study Chair — Montreal Children's Hospital of the MUHC; Melissa-Rosina Pasqua, M.D., Study Chair — Research Institute of the McGill University Health Centre
Locations (1):
- Research Institute of the McGill University Health Centre (RI-MUHC), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
After the completion of the trial, raw data will be shared for academic purposes upon request, according to the Materials Transfer Agreement.